CLINICAL TRIAL: NCT01448512
Title: University of Miami Developmental Center for AIDs Research Promoting Male Involvement to Improve PMTCT Uptake and Reduce Antenatal Infection
Brief Title: Promoting Male Involvement to Improve Prevention of Mother to Child Transmission (PMTCT) Uptake and Reduce Antenatal Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Deborah Jones, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 5P30AI073961-S; P30AI073961 (NIH)
Record Dates: First submitted 2011-09-26; First posted 2011-10-07 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: HIV; Pregnancy
Keywords: HIV; Pregnancy; Prevention; Couples
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Other): Participation in 4 time matched sessions on health education topics
  Interventions: Other: Usual Care
- PartnerPlus intervention (Experimental): Four group counseling sessions focused on prevention of mother to child transmission (PMTCT) sexual risk reduction & adherence.
  Interventions: Behavioral: PartnerPlus Intervention

INTERVENTIONS:
Behavioral: PartnerPlus Intervention — The intervention employs a closed, structured, group intervention limited to 10 participants (women or men). Four weekly, 11/2-2 hour sessions are led by a trained gender-congruent counselor and a peer facilitator and emphasize group participation, cognitive-behavioral skill building, sexual negotiation and experimentation with products.
  Other Names: Cognitive behavioral risk reduction intervention
  Arms: PartnerPlus intervention
Other: Usual Care — 4 time matched sessions focused on health education
  Other Names: Standard of Care
  Arms: Usual Care

SUMMARY:
This study will evaluate the impact of combining two evidence-based interventions: a couples risk reduction intervention with an evidence based medication adherence intervention designed to enhance male participation in combination with improving medication and prevention of mother to child transmission (PMTCT) adherence in antenatal clinics (ANCs). Clinics will be randomly assigned to experimental and control conditions and effectiveness of the combined intervention to enhance PMTCT as well as reduce antenatal seroconversion by both individuals and clinics will be examined. It is hypothesized that community clinics implementing PartnerPlus will have more effective PMTCT program adherence, as measured by total participant 1) maternal and paternal ANC and PartnerPlus visits, 2) maternal and paternal human immunodeficiency virus (HIV) Counseling & Testing (HCT) uptake, 3) maternal and infant antiretroviral (ARV) prophylaxis uptake, 4) maternal highly active antiretroviral therapy (HAART) uptake, 5) infant polymerase chain reaction (PCR) for HIV, and 5) maternal and infant HIV serostatus and that community clinics implementing PartnerPlus will have reduced sexual risk behavior, as measured by participant sexual barrier use.

DETAILED DESCRIPTION:
This study is a group-randomized controlled trial using a 2 x 6 comparison (Clinic, Experimental, Control x Time, Baseline, Post-Intervention, Pre-delivery 32 weeks, Pre-delivery day, Delivery, Post Partum). Twelve community health centers (CHCs) in communities within the Gert Sibande and Nkangala Districts in Mpumalanga, South Africa (SA) will be randomly assigned to condition in a 1:1 ratio. Six usual care condition clinics will provide the standard of care, PMTCT; six experimental condition clinics will offer PartnerPlus to mothers completing HIV testing, regardless of serostatus, who are willing to enroll with their male partners and participate in the integrated PartnerPlus intervention. This study will recruit 240 couples (n = 480 individuals); community clinics will recruit 2 cohort per clinic over 3 months (10 couples per cohort, n = 40, 120 individuals per condition).

ELIGIBILITY:
Inclusion Criteria:

* pregnant women age 18 and older who have received HCT (HIC Counseling & Testing) at the antenatal clinic (ANC),
* willing to attend PartnerPlus or prevention of mother to child transmission (PMTCT) visits with their male partners,
* male partners must also be available to participate and
* both partners must be willing to participate in the study.
* All participants will be current adult residents of Mpumalanga Province and agree to be attend four group sessions, 2 psychosocial assessments and 1 three day post-delivery assessment (maternal and infant blood sample).

Exclusion Criteria:

* Single mothers not being tested for HIV at the ANC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in number of ANC visits by mother and father from baseline to one month post intervention to 32 weeks to 3 days post partum | Baseline, one month, 32 weeks, 3 days post partum

SECONDARY OUTCOMES:
Change in Mother, father, infant HIV VCT from baseline to one month to 3 days post partum | Baseline, one month, 3 days post partum
Mother and infant ARV prophylaxis | 3 days post partum
Change in Maternal PMTCT ARV uptake from baseline to 32 weeks to 3 days post partum | Baseline, 32 weeks, 3 days post partum
Infant PCR | 6 weeks
Change in rate of condom use from baseline to one month to 3 days post partum | Baseline, one month, 3 days post partum

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peltzer, PhD, Study Director — Human Sciences Research Council; Deborah Jones, PhD, Principal Investigator — University of Miami
Locations (1):
- Human Sciences Research Council, Pretoria, Gauteng, South Africa